CLINICAL TRIAL: NCT02201069
Title: My Health Coach Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Zora Djuric, Research Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00087322
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Health Behavior
Keywords: nutrition; physical activity; sleep; weight loss
MeSH Terms: conditions — Health Behavior; Motor Activity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- health coaching (Experimental): 12 weeks of health coaching using weekly contact in the first month and biweekly contacts in months 2-3.
  Interventions: Behavioral: health coaching

INTERVENTIONS:
Behavioral: health coaching

SUMMARY:
The "My Health Coach Study" seeks to determine if health coaching by a medical assistant can help patients have better sleep, a better diet, be more physically active or lose weight, according to the recommendation of their health care provider.

DETAILED DESCRIPTION:
The aim of the study is to determine whether medical assistants (MAs) can assist primary care providers to achieve healthier lifestyles via better sleep, food choices, weight loss and/or increased physical activity in their patients. The hypothesis driving this research is that health coaching can be done by existing medical support staff to facilitate healthy lifestyles in a primary care setting. Coaching can maximize the health of the patient population in a cost-effective way if the coaching service is integrated into primary care clinics with minimal capital investment at the outset. A major focus will be on behaviors associated with weight management since this is the most common health issue in the U.S. today. This method, if successful, should be easily adaptable to other health behaviors and in most any medical practice that seeks to improve the health of its patient base in a cost-effective way.

In order to achieve a change in health behaviors, and especially weight loss, regular follow-up contacts are needed. Previous research has shown health coaching to be effective, but this has utilized programs that "add on" to the existing clinic structure. This type of coaching model is difficult to sustain. Utilizing existing staff for health coaching is a method we propose to more fully integrate this service into primary care clinics.

ELIGIBILITY:
Inclusion Criteria:

* adults age 21 and over
* referred by primary care physician for health coaching
* have telephone for follow-up
* English speaking

Exclusion Criteria:

* pregnant or trying to become pregnant

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 weeks

SECONDARY OUTCOMES:
Diet quality | 12 weeks
  adherence to USDA recommendations
Physical activity | 12 weeks
  adherence to physical activity recommendations of 30 min/day of at least moderate activity.
Sleep | 12 weeks
  Better sleep habits

OTHER OUTCOMES:
Quality of Life | 12 weeks
  stress, fatigue, self-efficacy, motivation

CONTACTS AND LOCATIONS:
Locations (1):
- Briarwood Family Medicine, Ann Arbor, Michigan, United States